CLINICAL TRIAL: NCT01757106
Title: The Safety and Feasibility of Administering Xenon to Patients Undergoing Off-pump Coronary Artery Bypass Graft Surgery: a Pilot Study
Brief Title: Xenon in Off-pump Coronary Artery Bypass Graft Surgery
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Universitaire Ziekenhuizen KU Leuven (Other)
Responsible Party: Principal Investigator, prof Dr Steffen Rex, Prof. Dr., Universitaire Ziekenhuizen KU Leuven
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: SR052012; 2012-002316-12 (EudraCT Number)
Record Dates: First submitted 2012-12-03; First posted 2012-12-28 (Estimated); Last update posted 2014-03-26 (Estimated); Status verified 2014-03

CONDITIONS: Coronary Artery Disease; Anesthesia
Keywords: xenon anesthesia; sevoflurane anesthesia; off-pump coronary artery bypass graft surgery
MeSH Terms: conditions — Coronary Artery Disease | interventions — Xenon; Sevoflurane

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No

ARMS (2):
- Drug: Xenon (Experimental): gaseous anesthetic, dosage: 50-60% (v/v) in oxygen, continuous application during surgery
  Interventions: Drug: Xenon
- Drug: Sevoflurane (Active Comparator): inhalative anesthetic, dosage: 1.4% (v/v) in 50% oxygen/medical air , continuous application during surgery
  Interventions: Drug: sevoflurane

INTERVENTIONS:
Drug: Xenon — general anaesthesia with xenon 50-60% in oxygen (FiO2=0.4-0.5)
  Arms: Drug: Xenon
Drug: sevoflurane — general anesthesia with sevoflurane 1.4% in 50% oxygen/medical air
  Arms: Drug: Sevoflurane

SUMMARY:
Purpose of this study is to test whether xenon application during off-pump-coronary artery bypass (OPCAB)-surgery is safe and feasible.

DETAILED DESCRIPTION:
The investigators hypothesize that xenon application during OPCAB-surgery performs non-inferiorly to the administration of the established anaesthetic sevoflurane with regard to haemodynamic stability, respiratory function, and depth of anesthesia. The evaluation of the outcome will include several secondary parameters such as the incidence of post-operative cardiovascular and neurovascular events, the incidence of organ dysfunction and further adverse events.

This study will further function as a pilot study for the evaluation of the incidence of postoperative delirium (POD) following OPCAB-surgery and xenon treatment. POD is a common complication of cardiac surgery/anaesthesia and may significantly affect the patients' mortality and outcome. Xenon possesses neuroprotective and anti-inflammatory qualities that may directly interfere with the pathogenesis of POD, as well as reducing other factors of perioperative organ injury including cardiac complications. Xenon´s favourable pharmacokinetic properties further result in rapid clearance from the brain, reducing any residual anaesthetic effects that may predispose to POD.

ELIGIBILITY:
Inclusion Criteria:

* Patients with coronary artery disease scheduled for elective OPCAB- surgery
* Patients willing and able to complete the requirements of this study
* Ejection Fraction > 30%

Exclusion Criteria:

* Lack of informed consent
* Age < 18 years
* Pregnancy
* chronic obstructive pulmonary disease (COPD) GOLD > II
* Renal dysfunction defined as serum-creatinine > 1.5 mg/dl
* Acute coronary syndrome during the last 24 hours; haemodynamic instability, requirement of inotropic support
* Single vessel grafting
* Disabling neuropsychiatric disorders (severe dementia, Alzheimer's disease, schizophrenia, depression), history of stroke with residuals, significant stenosis of carotid arteries, increased intracranial pressure
* Hypersensitivity to the study medication
* Presumed uncooperativeness or legal incapacity

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 42 (Actual)
Dates: Start 2012-12; Primary Completion 2013-07 (Actual); Study Completion 2014-01 (Actual)

PRIMARY OUTCOMES:
Feasibility/Safety of xenon anesthesia | Intraoperatively
  assessed by: depth of anesthesia, perioperative hemodynamic profile, peripheral and arterial oxygen saturation

SECONDARY OUTCOMES:
Major adverse cardiac and cerebral events (MACCE) | up to six months after surgery
  death from any cause; perioperative myocardial infarction and stroke
Incidence and duration of postoperative delirium | up to five days after surgery
  assessed with the Confusion Assessment Method (CAM-ICU)

OTHER OUTCOMES:
Other secondary efficacy/safety measures | up to five days after surgery
  Perioperative blood loss
Other secondary efficacy/safety measures | up to five days after surgery
  Requirement for blood (product) transfusion
Other secondary efficacy/safety measures | until discharge from the hospital
  Duration of postoperative intensive care unit and hospital stay
Other secondary efficacy/safety measures | up to five days after surgery
  Severity of postoperative critical illness as indicated by the sequential organ failure assessment (SOFA) score
Other secondary efficacy/safety measures | up to five days after surgery
  Perioperative renal function assessed by serum-creatinine levels and calculated creatinine clearance
other secondary efficacy/safety measures | up to five days after surgery
  Severity of postoperative critical illness as indicated by the new simplified acute physiology score (SAPS II)

CONTACTS AND LOCATIONS:
Overall Officials: Steffen Rex, PhD, Principal Investigator — UZ Leuven
Locations (1):
- University Hospitals Leuven, Leuven, Belgium

REFERENCES:
- [Derived] Al Tmimi L, Van Hemelrijck J, Van de Velde M, Sergeant P, Meyns B, Missant C, Jochmans I, Poesen K, Coburn M, Rex S. Xenon anaesthesia for patients undergoing off-pump coronary artery bypass graft surgery: a prospective randomized controlled pilot trial. Br J Anaesth. 2015 Oct;115(4):550-9. doi: 10.1093/bja/aev303. PMID 26385664